CLINICAL TRIAL: NCT01846793
Title: Phase 3 Multicenter Prospective Open Label Clinical Safety Evaluation of Re-Injection of NX-1207 for the Treatment of BPH: Two Doses 1-8 Years Apart
Brief Title: Phase 3 Evaluation of Re-Injection of NX-1207 for the Treatment of Benign Prostatic Hyperplasia (BPH)(NX02-0022)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nymox Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NX02-0022
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Benign Prostatic Hyperplasia; BPH; Lower Urinary Tract Symptoms (LUTS); LUTS
Keywords: Benign prostatic hyperplasia; BPH; Lower urinary tract symptoms; LUTS; LUTS secondary to BPH; LUTS/BPH; Benign prostatic obstruction (BPO); BPO; Bladder outlet obstruction; BOO
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Urinary Bladder Neck Obstruction | interventions — fexapotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label Injection of NX-1207 (Experimental): Intraprostatic injection of 2.5 mg NX-1207
  Interventions: Drug: NX-1207

INTERVENTIONS:
Drug: NX-1207 — 2.5 mg NX-1207 in 10 mL saline vehicle

SUMMARY:
This study is designed to demonstrate the safety and efficacy of a second transrectal intraprostatic injection of NX-1207 given to subjects with Benign Prostatic Hyperplasia (BPH) who previously received an injection of NX-1207 in an earlier U.S. clinical trial of NX-1207.

ELIGIBILITY:
Inclusion Criteria:

* Be male aged 45 or older.
* Sign an informed consent form.
* Be in good health.
* Received NX-1207 in a previous completed study (other than NX02-0020) or received NX-1207 or placebo in a concurrent U.S. study (NX02-0017 and NX02-0018) and completed their V10 (365 day) visit.
* Have Prostate Gland Volume ≥ 25 mL (25 g).

Exclusion Criteria:

* Surgery or minimally invasive surgical therapy (MIST) for treatment of BPH after first NX-1207 injection
* Post-void residual urine volume > 200 mL
* Presence of a symptomatic median lobe of the prostate
* History of use of self-catheterization for urinary retention.
* Urinary retention in the previous 12 months.
* Prostatitis
* Urinary tract infection more than once in the past 12 months
* Prostate or bladder cancer.
* Prostate-Specific Antigen (PSA) ≥ 10 ng/mL
* Poorly controlled diabetes
* History or evidence of illness or condition that may interfere with study or endanger subject
* Participation in a study of any investigational drug (other than NX-1207) or investigational device within the previous 90 days
* Use of specific prescribed medications that may interfere with study or endanger subject

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety | 180 days
  Safety parameters as determined by Adverse Events, clinical laboratory test results, vital signs, physical exam and electrocardiogram (ECG).

SECONDARY OUTCOMES:
Symptomatic Improvement | 90 days
  Symptomatic improvement as measured by the change in American Urological Association (AUA) Symptom Index from baseline at 90 days. The AUA Symptom Index is a standardized questionnaire that uses seven questions relating to associated BPH symptoms to provide an assessment of symptom severity on a scale from 0 (no symptoms) to 35 (most severe).
Prostate Volume Change | 90 days
  Change in prostate volume from baseline to 90 days as measured by transrectal ultrasonography
Change in Urinary Peak Flow | 90 days.
  Change in Urinary Peak Flow (Qmax) from baseline to 90 days as determined by urinary flow-rate recording (uroflowmetry).
Symptomatic Improvement | 180 days
  Symptomatic improvement as measured by the change in AUA Symptom Index from baseline at 180 days.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Laguna Beach, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., San Diego, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Aventura, Florida
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Naples, Florida
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Meridian, Idaho
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Jeffersonville, Indiana
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Shreveport, Louisiana
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Annapolis, Maryland
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Baltimore, Maryland
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Glen Burnie, Maryland
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Towson, Maryland
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Missoula, Montana
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Brick, New Jersey
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Garden City, New York
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., New York, New York
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Columbus, Ohio
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Dallas, Texas